CLINICAL TRIAL: NCT07145775
Title: Dexmedetomidine-esketamine-ropivacaine Versus Sufentanil-ropivacaine Combination for Epidural Labor Analgesia and Neonatal Outcomes: a Pilot Randomized Trial
Brief Title: Dexmedetomidine-esketamine-ropivacaine Versus Sufentanil-ropivacaine for Epidural Labor Analgesia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025R0269
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Epidural Analgesia; Labor Pain; Sufentanil; Dexmedetomidine; Esketamine; Ropivacaine
Keywords: epidural anagelsia; labor pain; sufentanil; dexmedetomidine; esketamine; ropivacaine
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: a randomized, double-blind, pilot trial with three parallel-arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Active Comparator): Epidural analgesia will be conducted with the sufentanil-ropivacaine combination (0.4 microgram/ml sufentanil + 0.072% ropivacaine; 100 microgram sufentanil + 18 ml 1% ropivacaine, diluted with normal saline to 250 ml).
  Interventions: Drug: sufentanil-ropivacaine combination
- experimental group 1 (Experimental): Epidural analgesia will be conducted with the dexmedetomidine-esketamine-ropivacaine combination 1 (0.4 microgram/ml dexmedetomidine + 0.15 mg/ml esketamine + 0.036% ropivacaine; 100 microgram dexmedetomidine + 37.5 mg esketamine + 9 ml 1% ropivacaine, diluted with normal saline to 250 ml).
  Interventions: Drug: dexmedetomidine-esketamine-ropivacaine combination 1
- experimental group 2 (Experimental): Epidural analgesia will be conducted with the dexmedetomidine-esketamine-ropivacaine combination 2 (0.4 microgram/ml dexmedetomidine + 0.2 mg/ml esketamine + 0.036% ropivacaine; 100 microgram dexmedetomidine + 50 mg esketamine + 9 ml 1% ropivacaine, diluted with normal saline to 250 ml).
  Interventions: Drug: dexmedetomidine-esketamine-ropivacaine combination 2

INTERVENTIONS:
Drug: sufentanil-ropivacaine combination — Epidural labor analgesia will be conducted using the sufentanil-ropivacaine combination (0.4 microgram/ml sufentanil + 0.072% ropivacaine).
  Other Names: epidural analgesia using the sufentanil-ropivacaine combination
  Arms: control group
Drug: dexmedetomidine-esketamine-ropivacaine combination 1 — Epidural labor analgesia will be conducted using the dexmedetomidine-esketamine-ropivacaine combination 1 (0.4 microgram/ml dexmedetomidine + 0.15 mg/ml esketamine + 0.036% ropivacaine).
  Other Names: epidural analgesia using the dexmedetomidine-esketamine-ropivacaine combination 1
  Arms: experimental group 1
Drug: dexmedetomidine-esketamine-ropivacaine combination 2 — Epidural labor analgesia will be conducted using the dexmedetomidine-esketamine-ropivacaine combination 2 (0.4 microgram/ml dexmedetomidine + 0.2 mg/ml esketamine + 0.036% ropivacaine).
  Other Names: epidural analgesia using the dexmedetomidine-esketamine-ropivacaine combination 2
  Arms: experimental group 2

SUMMARY:
Sufentanil-ropivacaine combination is commonly used for epidural labor anesthesia, but is associated with some adverse events. Dexmedetomidine and esketamine, each has been effectively used for neuraxial anesthesia in combination with local anesthetics. Plenty of evidences show that both dexmedetomidine and esketamine, combined with ropivacaine, are also effective as the sufentanil-ropivacaine combination when used for epidural labor analgesia. This pilot trial is designed to evaluate the efficacy and safety of the dexmedetomidine-esketamine-ropivacaine versus sufentanil-ropivacaine combination for epidural labor analgesia, and to test the feasibility of a future large randomized trial.

DETAILED DESCRIPTION:
Sufentanil-ropivacaine combination is commonly used for epidural labor anesthesia, but is associated with some adverse events. Dexmedetomidine and esketamine, each has been effectively used for neuraxial anesthesia in combination with local anesthetics. Plenty of evidences show that both dexmedetomidine and esketamine, combined with ropivacaine, are also effective as the sufentanil-ropivacaine combination when used for epidural labor analgesia.

The investigators hypothesize that the dexmedetomidine-esketamine-ropivacaine combination, by avoiding sufentanil and decreasing ropivacaine concentration, may provide non-inferior analgesia with less harmful effect on neonatal outcomes when compared with the sufentanil-ropivacaine combination. This pilot trial is designed to evaluate the efficacy and safety of the dexmedetomidine-esketamine-ropivacaine versus sufentanil-ropivacaine combination for epidural labor analgesia, and to test the feasibility of a future large randomized trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or above;
2. Single term cephalic pregnancy preparing for vaginal delivery;
3. Agreed to receive epidural labor analgesia.

Exclusion Criteria:

1. History of schizophrenia or epilepsy;
2. Presence of contraindications for epidural analgesia, including: (1) history of infectious disease of the central nervous system (poliomyelitis, cerebrospinal meningitis, encephalitis, etc.); (2) history of spinal or intra-spinal disease (trauma or surgery of spinal column, intra-spinal canal mass, etc.); (3) systemic infection (sepsis); (4) skin or soft tissue infection at the site of epidural puncture; (5) coagulopathy.
3. Relative contraindications for the use of dexmedetomidine, including prenatal bradycardia (HR<60 beats per minute) and second-degree or higher atrioventricular block;
4. Relative contraindications for the use of esketamine, including uncontrolled hypertension (systolic blood pressure >180 mmHg) and hyperthyroidism;
5. Not well controlled systemic diseases, including heart disease, liver disease, kidney disease, or an ASA classification >III;
6. Other conditions that are considered unsuitable for study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women preparing for vaginal delivery.
Enrollment: 300 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Time-weighted average score of pain intensity during labor | From start of analgesia to 2 hours after childbirth
  Pain intensity will be assessed with the numeric rating scale (an 11-point scale where 0=no pain and 10=the worst pain) at the fllowing timepoints: before analgesia, 10 and 30 minutes after loading dose, every hour during labor, full cervical dilation, immedlately after childbirth, and 2 hours after childbirth. Time-weighted average score will be calculated by summarizing the product of time interval between two adjacent pain scores multiplied by the average of corresponding pain scores, and then divided by the duration of epidural analgesia.

SECONDARY OUTCOMES:
Incidence of a composite of neonatal morbility | From immediate childbirth to 24 hours after childbirth
  Neonatal morbidity includes occurrence of any of the following events: 1-minute Apgar score <7, 5-minute Apgar score <7, neonatal umbilical artery blood gas PH<7.1, need for immediate assisted ventilation after birth, or admission to the neonatal ward or neonatal intensive care unit within 24 hours after birth.
Dosage of epidural labor analgesics | From start of analgesia to end of third stage or childbirth
  Including number of demanded boluses, number of delivered boluses, total volume, and hourly volume.
Incidence of persistent pain at 42 days postpartum | At 42 days postpartum
  Defined as a numeric rating scale of pain (an 11-point scale where 0=no pain and 10=the worst pain) at rest of 1 point or higher that persisted since childbirth.
Incidence of depression at 42 days postpartum | At 42 days postpartum
  Depression will be assessed with the Edinburgh Postnatal Depression Scale (EPDS; score range 0-30, with higher score indicating more severe depression). An Edinburgh depression score of 10 points or higher indicates presence of depressive symptoms.

OTHER OUTCOMES:
Scores of pain intensity at various timepoints during labor | Up to 2 hours after childbirth
  Pain intensity will be assessed with the numeric rating scale (an 11-point scale where 0=no pain and 10=the worst pain) at the fllowing timepoints: before analgesia, 10 and 30 minutes after loading dose, every hour during labor, full cervical dilation, immedlately after childbirth, and 2 hours after childbirth.
Scores of sedation at various timepoints during labor | Up to 2 hours after childbirth
  Maternal sedation will be assessed with the Ramsay Agitation-Sedation Scale (1=anxious and agitated or restless; 2=awake, quiet and cooperative; 3=drowsy but responding to verbal commands; 4=lightly asleep but responding to touch or pain; 5=asleep but slowly responding to touch or pain; 6=deeply asleep and does not respond) at the fllowing timepoints: before analgesia, 10 and 30 minutes after loading dose, every hour during labor, full cervical dilation, immedlately after childbirth, and 2 hours after childbirth.
Degree of lower limb motor block at various timepoints during labor | Up to 2 hours after childbirth
  Lower limb motor block will be assessed with the modified Bromage scale (0=no motor loss; 1=inability to flex the hip; 2=inability to flex the knee; 3=inability to flex the ankles) at the fllowing timepoints: before analgesia, 10 and 30 minutes after loading dose, every hour during labor, full cervical dilation, immedlately after childbirth, and 2 hours after childbirth.
Duration of each stage of labor | From start of labor to end of third stage
  Including durations of the first, second, and third stages of labor.
Mode of delivery | From start of labor to childbirth
  Mode of delivery
Subjective sleep quality during the first night after childbirth | Up to 24 hours after childbirth
  Subjective sleep quality will be assessed with the numeric rating scale (an 11-point scale where 0=the best sleep and 10=the worst sleep) in the first morning after childbirth.
Time to breastfeeding | Up to 24 hours after childbirth
  Time to breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lou S, Du Q, Yu L, Wang Q, Yu J, Mei Z. ED90 of epidural esketamine with 0.075% ropivacaine for labor analgesia in nulliparous parturients: a prospective, randomized and dose-finding study. Front Pharmacol. 2023 May 5;14:1169415. doi: 10.3389/fphar.2023.1169415. eCollection 2023. PMID 37214452
- [Result] Zhang Y, Cui F, Ma JH, Wang DX. Mini-dose esketamine-dexmedetomidine combination to supplement analgesia for patients after scoliosis correction surgery: a double-blind randomised trial. Br J Anaesth. 2023 Aug;131(2):385-396. doi: 10.1016/j.bja.2023.05.001. Epub 2023 Jun 9. PMID 37302963
- [Result] Li K, Chai Z, Deng C, Niu G, Geng X, Zhang Y, Wang Y, Wang T. Effects of epidural esketamine versus sufentanil on labor analgesia and postpartum depression: a retrospective cohort study. BMC Anesthesiol. 2025 Jan 7;25(1):6. doi: 10.1186/s12871-024-02846-6. PMID 39773190
- [Result] Xu L, Li S, Zhang C, Zhou Y, Chen X. Esketamine administered epidurally as an adjuvant to epidural ropivacaine for labour analgesia: a prospective, double-blind dose-response study. BMJ Open. 2024 Nov 2;14(11):e071818. doi: 10.1136/bmjopen-2023-071818. PMID 39488417
- [Result] Richards ND, Howell SJ, Bellamy MC, Beck J. The diverse effects of ketamine, jack-of-all-trades: a narrative review. Br J Anaesth. 2025 Mar;134(3):649-661. doi: 10.1016/j.bja.2024.11.018. Epub 2025 Jan 2. PMID 39753406
- [Result] Jin KX, Deng CM, Ding T, Qu Y, Wang DX. Impact of dexmedetomidine-ropivacaine versus sufentanil-ropivacaine combination for epidural labour analgesia on neonatal outcomes: a pilot randomised clinical trial. BMJ Open. 2024 Dec 22;14(12):e090208. doi: 10.1136/bmjopen-2024-090208. PMID 39806707
- [Result] Qian M, Gao F, Liu J, Xu P. Dexmedetomidine versus fentanyl as adjuvants to ropivacaine for epidural anaesthesia: A systematic review and meta-analysis. Int J Clin Pract. 2021 May;75(5):e13772. doi: 10.1111/ijcp.13772. Epub 2020 Dec 20. PMID 33078536
- [Result] Rao S, Rajan N. Dexmedetomidine as an Adjunct for Regional Anesthetic Nerve Blocks. Curr Pain Headache Rep. 2021 Feb 3;25(2):8. doi: 10.1007/s11916-020-00926-z. PMID 33533982
- [Result] Armstrong S, Fernando R. Side Effects and Efficacy of Neuraxial Opioids in Pregnant Patients at Delivery: A Comprehensive Review. Drug Saf. 2016 May;39(5):381-99. doi: 10.1007/s40264-015-0386-5. PMID 26832926